CLINICAL TRIAL: NCT02723344
Title: Biological Signature and Safety of an Immunomodulatory Probiotic Intervention for Veterans With Co-Occurring Mild TBI and PTSD
Brief Title: Biological Signatures, Probiotic Among Those With mTBI and PTSD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: N2232-P
Record Dates: First submitted 2016-03-01; First posted 2016-03-30 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Mild Traumatic Brain Injury; Post Traumatic Stress Disorder
Keywords: PTSD; Mild TBI; Probiotic; Inflammation
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic; Inflammation

STUDY DESIGN:
Intervention Model Description: Biologic
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L. reuteri (Experimental): Commercially available L. reuteri (deposited in the Deutsche Sammlung von Mikroorganismen und Zellkulturen (DSMZ) and referenced as DSM 17938; Gerber Soothe Colic Drops, 100 million CFU/5 drops; formerly known as L. reuteri ATCC 55730) will be used in the proposed study. L. reuteri (phylum Firmicutes) is a gram-positive anaerobic commensal bacteria found in the gut microbiome of humans. Independent testing of the viability of the commercial product will be conducted in our laboratories by diluting drops, plating on agar in triplicate, and anaerobic culturing at 37 oC. The commercial strain (DSM 17938) has been used to improve intestinal functions in infants and reduce symptoms of infantile colic.
  Interventions: Dietary Supplement: of Lactobacillus reuteri (L. reuteri; DSM 17938)
- Sunflower and medium chain triglyceride oils (Placebo Comparator): Sunflower and medium chain triglyceride oils
  Interventions: Other: Sunflower and medium chain triglyceride oils

INTERVENTIONS:
Dietary Supplement: of Lactobacillus reuteri (L. reuteri; DSM 17938) — Commercially available L. reuteri (deposited in the Deutsche Sammlung von Mikroorganismen und Zellkulturen (DSMZ) and referenced as DSM 17938; Gerber Soothe Colic Drops, 100 million CFU/5 drops; formerly known as L. reuteri ATCC 55730) will be used in the proposed study. L. reuteri (phylum Firmicutes) is a gram-positive anaerobic commensal bacteria found in the gut microbiome of humans. Independent testing of the viability of the commercial product will be conducted in our laboratories by diluting drops, plating on agar in triplicate, and anaerobic culturing at 37 oC. The commercial strain (DSM 17938) has been used to improve intestinal functions in infants and reduce symptoms of infantile colic.
  Arms: L. reuteri
Other: Sunflower and medium chain triglyceride oils — Placebo
  Other Names: Placebo
  Arms: Sunflower and medium chain triglyceride oils

SUMMARY:
Exaggerated inflammation in the body and brain is thought to play a role in the vulnerability to and aggravation and perpetuation of adverse consequences among those with co-occurring mild TBI (mTBI) and post-traumatic stress disorder (PTSD). The proposed study begins the process of investigating the use of a natural immunoregulatory/anti-inflammatory probiotic to treat chronic symptoms associated with co-occurring mTBI and PTSD among Veterans. By looking at the impact of probiotic supplementation on biological signatures of increased inflammation, as reflected by the gut microbiota, gut permeability, and biomarkers of peripheral inflammation, this study may lead to the identification of a novel intervention for the treatment of symptoms associated with these frequently co-occurring conditions.

DETAILED DESCRIPTION:
United States military Veterans from recent conflicts are coping with symptoms related to mild traumatic brain injury (mTBI), persistent post concussive (PPC) symptoms, and posttraumatic stress disorder (PTSD). Many Veterans are resistant to conventional health and mental health interventions (e.g., medication, psychotherapy), and often symptoms are not significantly improved by traditional treatments. Moreover, there are limited treatments for symptoms associated with both conditions, which frequently co-occur. Alternative treatment methods are needed. One potential common underlying feature of both mTBI and PTSD is exaggerated inflammation, both peripherally and in the central nervous system, which is thought to play an important role in the vulnerability to, aggravation of, and perpetuation of adverse consequences of these often co-occurring conditions. Therefore, a novel intervention strategy would be the use of immunoregulatory/anti-inflammatory probiotics to reduce inflammation. In this study, the investigators will investigate the effects of an immunoregulatory probiotic on both biological signatures of systemic inflammatory processes and proximal signatures of probiotic administration. Lactobacillus reuteri (L. reuteri), a commensal organism that colonizes the human gut mucosa, suppresses mucosal inflammation via inhibition of the production of proinflammatory cytokines, and is the probiotic of interest. Specific aims of the study are to determine the: 1) effects of L. reuteri on biological signatures of gut microbiota, gut permeability, systemic inflammation processes, and stress responses; 2) feasibility of L. reuteri supplementation; 3) acceptability of L. reuteri supplementation; and 4) tolerability and safety of L. reuteri supplementation. Project aims will be assessed using a longitudinal, double blind, randomized placebo-controlled design. Participants will be Veterans with PPC symptoms, PTSD, and evidence of elevated systemic inflammation (based on high baseline plasma C-reactive protein [CRP] concentrations). After initial evaluation procedures, 20 participants will be randomized to probiotic supplementation and 20 will be randomized to placebo supplementation. The proposed line of research addresses the Office of Rehabilitation Research and Development (RR&D) Service's goal of identifying means of intervening to increase function among those with mTBI and co-occurring psychiatric conditions. Long-term, this study may lead to a paradigm shift in the manner by which the investigators target clinical symptoms associated with PPC and PTSD symptoms, by beginning the process of supporting a multitargeted, neuroprotective approach.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one deployment in support of Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF)/Operation New Dawn (OND)
* History of mTBI per the Ohio State University (OSU) TBI-ID85 with any endorsement of post concussive symptoms (PCS) associated with an mTBI, which occurred at least 6 months prior to the baseline assessment
* Current symptoms in 3 or more of the following ICD-10 Post Concussive Symptom86 categories as measured by the Rivermead Post Concussive Symptom Questionnaire (RPCSQ87; score of 2 or greater per symptom to qualify):

  * headache
  * dizziness
  * malaise
  * fatigue
  * noise intolerance
  * irritability
  * depression
  * anxiety
  * emotional lability
  * subjective concentration
  * memory
  * intellectual difficulties
  * and/or insomnia
* Current diagnosis of PTSD per the Clinician Administered PTSD Scale-5 (CAPS-5)88
* Medical clearance by study physicians to participate in the protocol
* Age between 18 and 50
* Ability to provide informed consent
* Willingness not to take probiotic supplements (pills, tablets, oils, etc.) other than the product provided in the clinical study until all study procedures are completed
* Willingness to provide blood, as well as stool samples

Exclusion Criteria:

* Inability to adequately respond to questions regarding the informed consent procedure
* Currently involved in the criminal justice system as a prisoner or ward of the state
* Non-English speaking
* Current (past month) alcohol or substance abuse or dependence
* Lifetime history of bipolar disorder or psychosis or anxiety disorders (excluding PTSD)
* Current major depressive disorder (MDD)
* Consistent (e.g., 5x/week or greater) probiotic supplementation within the last month, including probiotic food products such as yogurt, as determined by phone screen interview and Probiotic Food Check List
* Receiving antibiotics within the last month; use of topical antibiotics or topical steroids on the face, scalp, or neck or on arms, forearms, or hands within the previous 7 days
* Receiving medications that interfere with gut motility (opiates, loperamide, stool softeners)
* Presence of central venous catheters (CVCs)
* Gastrointestinal (GI) barriers as identified by the 2-week run-in period as determined by the study team (e.g., daily GI discomfort with frequent diarrhea prior to supplementation)
* Participation in conflicting interventional research protocol
* Body mass index (BMI) greater than or equal to 35 or less than or equal to 18
* Vital signs outside of acceptable range, i.e., blood pressure >160/100, oral temperature >100 F, pulse >100
* Use of any of the following drugs within the last 6 months:

  * systemic antibiotics
  * antifungals
  * antivirals or antiparasitics (intravenous, intramuscular, or oral)
  * oral
  * intravenous
  * intramuscular
  * nasal or inhaled corticosteroids
  * cytokines or cytokine inhibitors
  * methotrexate or immunosuppressive cytotoxic agents
* Acute disease at the time of enrollment (defer sampling until subject recovers)

  * Acute disease is defined as the presence of a moderate or severe illness with or without fever
* Chronic, clinically significant (unresolved, requiring on-going medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality, as determined by medical history or physical examination other than irritable bowel syndrome (IBS)
* History of cancer except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet
* Positive test for human immunodeficiency virus (HIV), Hepatitis B virus, or Hepatitis C virus
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection
* Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time
* Regular urinary incontinence necessitating use of incontinence protection garments
* Female who is pregnant or lactating
* Treatment for or suspicion of ever having had toxic shock syndrome
* Those receiving immunosuppressive drugs or treatment including antineoplastic therapy, post-transplantation immunosuppressive therapy, and/or radiation therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brenner LA, Forster JE, Stearns-Yoder KA, Stamper CE, Hoisington AJ, Brostow DP, Mealer M, Wortzel HS, Postolache TT, Lowry CA. Evaluation of an Immunomodulatory Probiotic Intervention for Veterans With Co-occurring Mild Traumatic Brain Injury and Posttraumatic Stress Disorder: A Pilot Study. Front Neurol. 2020 Oct 20;11:1015. doi: 10.3389/fneur.2020.01015. eCollection 2020. PMID 33192959
- See also: Click here for more information about this study: Biological Signature and Safety of an Immunomodulatory Probiotic Intervention for Veterans with Co-Occurring Mild TBI and PTSD — http://www.mirecc.va.gov/visn19/research/recruitment/index.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Although 75 participants were consented and enrolled in the study, 31 participants met inclusion criteria and continued participation.
Groups:
- Placebo: Allocated to Placebo
- L Reuteri: Allocated to L reuteri
Period: Overall Study
Arm/Group | Placebo | L Reuteri
Started | 15 | 16
Completed | 15 | 12
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Population: Prior to randomization
Groups:
- Placebo: Sham Probiotic
- L Reuteri: Probiotic
- Total: Total of all reporting groups
Arm/Group | Placebo | L Reuteri | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (6.2) | 37.9 (7.3) | 37.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 16 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 11 | 21
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: C-Reactive Protein Change
Description: Inflammation - Biological Signature (Blood)
Time Frame: Baseline and approximately 10 weeks
Population: A sufficient amount of plasma was not available to run CRP on 1 participant in the placebo group and 2 participants in the L reuteri group.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | L Reuteri
Number analyzed (Participants) | 14 | 10
mg/L | 0.113 (1.2) | -0.625 (1.1)
Statistical Analysis 1: Comparison: Placebo vs L Reuteri; Test type: Other; p = .056, Wilcoxon-rank sum

2. Secondary Outcome: Tumor Necrosis Factor Change
Description: Inflammation - Biological Signature (Blood)
Time Frame: 2 weeks and approximately 10 weeks
Population: A sufficient amount of plasma was not available to run TNF on 1 participant in the placebo group and 3 participants in the L reuteri group.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | L Reuteri
Number analyzed (Participants) | 14 | 9
pg/ml | -0.62 (1.4) | -2.1 (8.2)
Statistical Analysis 1: Comparison: Placebo vs L Reuteri; Test type: Other; p = .26, Wilcoxon (Mann-Whitney) — Wilcoxon Rank-Sum

3. Other Pre Specified Outcome: Visual Analog Scale
Description: The VAS was administered during the Trier Social Stress Task (TSST). The VAS is self-reported stress response on a Likert scale (1-10). A higher score indicates greater perceived stress. In the TSST, participants are asked to give a 5-minute speech and perform a math task. The VAS was administered at the baseline of the TSST, after the Speech Task, and after the Math Task.
Time Frame: Approximately 10 weeks
Population: VAS was administered at T3 therefore data was only available on participants who completed the study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | L Reuteri
Number analyzed (Participants) | 15 | 12
score on a scale
  TSST Baseline | 4.13 [2.77 to 5.50] | 5.38 [3.85 to 6.90]
  TSST After Speech | 5.29 [4.04 to 6.54] | 6.25 [4.87 to 7.63]
  TSST After Math | 6.44 [5.06 to 7.84] | 7.13 [5.60 to 8.65]

4. Other Pre Specified Outcome: Interleukin 6 Change
Description: Inflammation - Biological Signature (Blood)
Time Frame: 2 weeks and approximately 10 weeks
Population: A sufficient amount of plasma was not available to run IL6 on 1 participant in the placebo group and 3 participants in the L reuteri group.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | L Reuteri
Number analyzed (Participants) | 14 | 9
pg/ml | .22 (2.4) | -.07 (7.7)
Statistical Analysis 1: Comparison: Placebo vs L Reuteri; Test type: Other; p = .64, Wilcoxon Rank-Sum

5. Other Pre Specified Outcome: Interleukin 10 Change
Description: Inflammation - Biological Signature (Blood)
Time Frame: 2 weeks and approximately 10 weeks
Population: A sufficient amount of plasma was not available to run IL10 on 1 participant in the placebo group and 3 participants in the L reuteri group.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | L Reuteri
Number analyzed (Participants) | 14 | 9
pg/ml | 0.15 (0.85) | -0.23 (2.0)

6. Other Pre Specified Outcome: Intestinal Fatty Acid Binding Protein (IFABP) Change
Description: Gut Permeability (Blood) - IFABP, measured by ELISA
Time Frame: 2 weeks and approximately 10 weeks
Population: A sufficient amount of plasma was not available to run IFABP on 3 participants in the placebo group and 2 participants in the L reuteri group.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | L Reuteri
Number analyzed (Participants) | 12 | 10
pg/ml | -0.09 (0.45) | -0.04 (0.16)

7. Other Pre Specified Outcome: D-amino Acid Oxidase (DAO) Change
Description: Gut Permeability (Blood) - DAO, measured by ELISA
Time Frame: 2 weeks and approximately 10 weeks
Population: A sufficient amount of plasma was not available to run DAO on 5 participants in the placebo group and 4 participants in the L reuteri group.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | L Reuteri
Number analyzed (Participants) | 10 | 8
pg/ml | -0.11 (0.24) | 0.03 (0.12)

8. Other Pre Specified Outcome: Generic Assessment of Side Effects-Probiotics (GASE-P)
Description: This measure of tolerability consists of 36 symptom descriptions organized by body parts. Participants are asked to rate if these symptoms were either "not present", "mild", "moderate", or "severe" in the past week related to supplementation. Total severity scores range 0-108. A higher severity score indicates more symptom severity. Total symptom scores range 0-36. A higher symptom score indicates more symptoms.
Time Frame: Time 1 (Baseline), Time 2 (2 weeks), and Time 3 (10 weeks)
Population: 2 participants in the L reuteri group were lost to follow at Time 2, and then 2 more participants were lost to follow at Time 3.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | L Reuteri
Number analyzed (Participants) | 15 | 16
score on a scale
  Time 1 - Severity | 25.6 (13.9) | 28.1 (12.7)
  Time 1 - Symptom Count | 14.4 (5.5) | 15.9 (6.4)
  Time 2 - Severity: number analyzed (Participants) | 15 | 14
  Time 2 - Severity | 22.1 (13.2) | 23.7 (8.8)
  Time 2 - Symptom Count: number analyzed (Participants) | 15 | 14
  Time 2 - Symptom Count | 12.4 (6.4) | 15.6 (4.8)
  Time 3 - Severity: number analyzed (Participants) | 15 | 12
  Time 3 - Severity | 11.7 (11.3) | 14.3 (12.0)
  Time 3 - Symptom Count: number analyzed (Participants) | 15 | 12
  Time 3 - Symptom Count | 6.5 (4.5) | 9.8 (8.5)

ADVERSE EVENTS:
Time Frame: Through study competition, an average of 10 weeks
Arm/Group | Placebo | L Reuteri
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02723344/Prot_SAP_000.pdf